CLINICAL TRIAL: NCT02064049
Title: A Pilot Study to Assess the Feasibility of Hepatitis C Virus (HCV) Treatment as Prevention With Interferon-free Direct Acting Antivirals (DAAs) in the Prison Setting
Brief Title: Surveillance and Treatment of Prisoners With Hepatitis C
Acronym: SToP-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1302
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; People who inject drugs; Drug users; Direct acting antiviral (DAA); Infectious diseases; Prisoners
MeSH Terms: conditions — Hepatitis C; Drug Misuse; Communicable Diseases | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatitis C treatment (Experimental): All prisoners (in participating correctional centres) with hepatitis c, as identified during the hepatitis C surveillance phase of the study will be offered treatment for hepatitis C. The treatment course is sofosbuvir/velpatasvir 400/100mg for 12 weeks (1 tablet once daily).
  Interventions: Drug: Sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: Sofosbuvir/velpatasvir — The treatment phase will commence in year 2. This is 12 weeks of the pangenotypic sofosbuvir/velpatasvir 400/100mg, coformulated into one tablet daily.
  Other Names: Epslusa

SUMMARY:
The purpose of the study is to assess how feasible it is to treat and prevent the transmission of Hepatitis C in the prison setting to achieve substantial reductions in the incidence and prevalence of Hepatitis C.

It is hypothesised that a rapid scale-up of Hepatitis C Virus (HCV) treatment with interferon-free Direct Acting Anti-virals (DAAs) in prison inmates will achieve a >50% reduction in the incidence of HCV infection over a two year period in the prison setting.

DETAILED DESCRIPTION:
The study will be conducted initially in two maximum security prisons located in New South Wales, Australia and comprises four phases:

Phase 1, Surveillance of HCV Incidence and Prevalence and Liver Disease Burden:

The HCV incidence and prevalence phase is a prospective longitudinal cohort. HCV incidence and prevalence and liver disease burden will be monitored through regular six-monthly cross-sectional surveys of participants for 3.5 years.

Phase 2, Modelling:

The data from year 1 of the surveillance of HCV incidence and prevalence phase will be used to model the number of participants required to be treated to demonstrate a 50% reduction in incidence.

Phase 3, Treatment Intervention:

The treatment intervention will only be conducted in one of the maximum security prisons (Treatment Prison). The second prison will continue to care for HCV infected inmates as per standard of care (Control Prison). The intervention component of this study will consist of a phase IV open-label study of interferon-free DAAs for the treatment of HCV infection. The treatment phase will commence in year 2 and will be two years in duration. The exact drug combination and regimen to be used in the treatment intervention will be determined in year 1 once phase II and III data of sofosbuvir and ledipasvir and other potential interferon-free DAA regimens are published. The exact number of participants required to demonstrate a 50% reduction in incidence will be determined during the modelling phase.

Phase 4, Cost-effectiveness:

During the treatment intervention phase participants will be required to complete a survey to obtain estimates of health outcomes (EQ-5D survey) at regular intervals. This data will be used by the health economist to determine the cost effectiveness of treatment as prevention in the prison setting.

ELIGIBILITY:
Surveillance of HCV Incidence and Prevalence Inclusion criteria

1. 18 years of age or older
2. Voluntarily signed the (surveillance phase) informed consent form.
3. Adequate English and mental health status to provide written informed consent and comply with study procedures

Exclusion criteria

1) Prisoners of a security classification which makes clinic attendance for study visits logistically difficult 5.2 Treatment Intervention Inclusion criteria

1. 18 years of age or older.
2. Voluntarily signed the (treatment phase) informed consent form.
3. Detectable HCV RNA in plasma.
4. HCV genotypes 1-6
5. Anticipated incarceration duration >12 weeks following the planned commencement of therapy.
6. Compensated liver disease where the following criteria must be met:

   1. INR< 1.8
   2. Albumin >30 g/L
   3. Bilirubin <35umol/L
7. Prisoners with Fibroscan > 12KPa or AFP >50 ng/mL must have an abdominal ultrasound or CT scan without evidence of hepatocellular carcinoma within 2 months prior to screening.
8. Negative pregnancy test at baseline (females of childbearing potential only).
9. [For prisoners released during treatment or follow-up] If engaging in sexual intercourse which may potentially result in pregnancy, all fertile males must be using effective contraception during treatment and during the 90 days after treatment end, and all fertile females must be using effective contraception during treatment and during the 30 days after treatment end
10. If co-infection with HIV is documented, the subject must meet the following criteria:

    1. Antiretroviral (ARV) untreated for >8 weeks preceding screening visit with CD4 T cell count >500 cells/mm3 OR
    2. On a stable ARV regimen for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and an undetectable plasma HIV RNA level.

       * Suitable ARV include:

         * Nucleos(t)ide reverse transcriptase inhibitors: Tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), emtricitabine (FTC)Non-nucleoside reverse transcriptase inhibitors: Rilpivirine
         * Protease inhibitors: Atazanavir, darunavir, lopinavir, ritonavir
         * Integrase inhibitors: Dolutegravir, raltegravir, elvitegravir/cobicistat
       * Contraindicated ARV include:

         * Efavirenz (50% reduction in velpatasvir exposure)
         * Didanosine
         * Zidovudine
         * Tipranavir Other ARV agents may be permissible at the time of study commencement pending further drug-drug interaction studies; please discuss with the Medical Monitor.

Exclusion criteria

1. Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) <6 months prior to the first dose of study drug.
2. Any investigational drug <6 weeks prior to the first dose of study drug.
3. History or other evidence of clinical hepatic decompensation (i.e. ascites, encephalopathy or oesophageal variceal haemorrhage)
4. Solid organ transplant
5. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the prisoner treatment, assessment or compliance with the protocol; prisoners currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded.
6. History of any of the following:

   1. Malignancy within 5 years prior to screening, with exception of specific cancers that may have been cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are also excluded.
   2. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
7. Any of the following lab parameters at screening:

   1. ALT > 10 x ULN
   2. AST > 10 x ULN
   3. Direct bilirubin > 1.5 x ULN
   4. Platelets < 50,000/uL
   5. Creatinine clearance < 60 mL/min
   6. Haemoglobin < 11 g/dL for females ; < 12 g/dL for males
   7. Albumin < 30g/L
   8. INR > 1.5 ULN unless subject has known haemophilia or is stable on an anticoagulant regimen affecting INR
8. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day)
9. Known hypersensitivity to VEL, SOF or formulation excipients.
10. Use of prohibited concomitant medications as described in section 6.2
11. Pregnant or nursing female
12. Ongoing severe psychiatric disease as judged by the treating physician.
13. Frequent injecting drug use that is judged by the treating physician to compromise treatment safety.
14. Inability or unwillingness to provide informed consent or abide by the requirements of the study.
15. Any other criteria that is judged by the treating physician to potentially compromise treatment safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3692 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Hepatitis C virus (HCV) incidence | 2 years
  Incidence of HCV infection over a two year period in a network of four participating correctional centres.

SECONDARY OUTCOMES:
Hepatitis C virus prevalence | 2 years
  Change in prevalence of HCV infection over a two year period in a network of four participating correctional centres.
SVR12 | 24 weeks
  The proportion of patients with undetectable HCV RNA at 12 weeks following the end of treatment (SVR12)
ETR | 12 weeks
  The proportion of patients with an end of treatment response (ETR)
Rapid Virological Response (RVR) | 4 weeks
  The proportion of patients with undetectable HCV RNA at 4 weeks following the initiation of treatment (RVR)
Treatment adherence | 12 weeks
  The proportion adherent to therapy (both on-treatment adherence and treatment discontinuation) and the association between adherence and response to treatment
Number of patients with adverse events | 16 weeks
  Safety and tolerability of the treatment regimen
Treatment uptake | 2 years
  The rate of HCV treatment uptake among eligible inmates and reasons for non-uptake
On-treatment change in illicit drug use | 24 weeks
  Changes in illicit drug use behaviours during treatment
HCV reinfection rate | 2 years
  The rate of HCV reinfection following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Dore, MBBS,PhD, Principal Investigator — Kirby Institute, University of New South Wales; St Vincent's Hospital Sydney
Locations (4):
- Australia (4):
  - Goulburn Correctional Centre, Goulburn, New South Wales
  - Lithgow Correctional Centre, Lithgow, New South Wales
  - Dillwynia Correctional Centre, Windsor, New South Wales
  - Outer Metropolitan Multipurpose Correctional Centre, Windsor, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shih STF, Stone J, Martin NK, Hajarizadeh B, Cunningham EB, Kwon JA, McGrath C, Grant L, Grebely J, Dore GJ, Lloyd AR, Vickerman P, Chambers GM. Scale-up of Direct-Acting Antiviral Treatment in Prisons Is Both Cost-effective and Key to Hepatitis C Virus Elimination. Open Forum Infect Dis. 2023 Dec 18;11(2):ofad637. doi: 10.1093/ofid/ofad637. eCollection 2024 Feb. PMID 38344130
- [Derived] Carson JM, Dore GJ, Lloyd AR, Grebely J, Byrne M, Cunningham E, Amin J, Vickerman P, Martin NK, Treloar C, Martinello M, Matthews GV, Hajarizadeh B; Surveillance and Treatment of Prisoners With Hepatitis C (SToP-C) Study Group. Hepatitis C Virus Reinfection Following Direct-Acting Antiviral Treatment in the Prison Setting: The SToP-C Study. Clin Infect Dis. 2022 Nov 14;75(10):1809-1819. doi: 10.1093/cid/ciac246. PMID 35362522
- [Derived] Hajarizadeh B, Grebely J, Byrne M, Marks P, Amin J, McManus H, Butler T, Cunningham EB, Vickerman P, Martin NK, McHutchison JG, Brainard DM, Treloar C, Chambers GM, Grant L, Mcgrath C, Lloyd AR, Dore GJ; SToP-C study group. Evaluation of hepatitis C treatment-as-prevention within Australian prisons (SToP-C): a prospective cohort study. Lancet Gastroenterol Hepatol. 2021 Jul;6(7):533-546. doi: 10.1016/S2468-1253(21)00077-7. Epub 2021 May 7. PMID 33965006